CLINICAL TRIAL: NCT05988645
Title: Performance and Safety of MiWEndo-assisted Colonoscopy: MiWEndo II (Pivotal Study)
Brief Title: Performance and Safety of MiWEndo-assisted Colonoscopy (MiWEndo II)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MiWEndo Solutions S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MW II-CIP
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Colorectal Polyp; Colorectal Adenoma; Colorectal Adenomatous Polyp; Colorectal Adenocarcinoma; Colorectal Neoplasms
Keywords: microwave imaging; colonoscopy; early diagnosis; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Traditional safety and performance study, following a single-center prospective and noncomparative.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MiWEndo + colonoscope (Experimental): All patients will be explored with MiWEndo as an accessory to colonoscopy
  Interventions: Device: MiWEndo System

INTERVENTIONS:
Device: MiWEndo System — All colonoscopies will be performed with high-definition technology. The MiWEndo System will be fitted to the tip of the endoscope before colonoscopy is started and connected to the microwave processor unit. Endoscopies will be performed by experienced endoscopists who will be previously trained on the use of the MiWEndo System. The MiWEndo Analyzer will be managed by the assistant.
  At the beginning of the extubation, the MiWEndo System will be turned on and the endoscopist will put music headphones on (blind to the results of MiWEndo).
  In case one of them identifies a polyp, the exploration will be stopped and check if it has been detected by the alternative method as well. All the polyps will be resected and sent to the Pathological Department for histological analysis following the usual clinical practice. A stopwatch will be used to measure both total procedure time and withdrawal time.

SUMMARY:
The study involves the planned use of a new microwave-based device during colonoscopy procedures in 50 patients to assess the performance and safety of its use for detection of colorectal polyps and lack of normal clinical practice modification. The device is a final design version, which has been previously tested in several preclinical studies (including phantom studies, an ex vivo study with human tissues, and an in vivo study with porcine model) and in a pilot study in humans (NCT05477836)

DETAILED DESCRIPTION:
This study is designed as a single-center prospective, non-comparative study in 50 patients, whereby data will be subject to an analytical description, rather than to a statistical treatment (refer to Statistical design and analysis).

In this study the principal aims are to assess the performance and safety of the device for the detection of colorectal polyps when used as an accessory to colonoscopy. Relevant claims to verify in this study are that the device will detect in first instance polyps not detected initially with the endoscopic image and can be used without ADEs, without any change in the current clinical practice, as well as without any major difficulty by the endoscopist, neither in the preparation nor in the use of the device during exploration.

In addition, in the first phase of the study (n=15 patients), the study aims to gather real clinical data with the use of the device to optimise the processing software that will be key to demonstrate MiWEndo's performance on the second part of the study (n=35 patients).

Consequently, principal and secondary objectives of this investigation, are:

Principal objectives:

* To assess the performance of MiWEndo-assisted colonoscopy in the detection of colorectal polyps.
* To assess the safety of MiWEndo-assisted colonoscopy.

Secondary objectives:

* To assess the perception of difficulty by the endoscopist when the device is used.
* To provide exploratory analysis of differences in MiWEndo-assisted colonoscopy in different groups of patients to guide future RCT.
* To assess the patient's comfort.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a previously detected polyp in the rectum referred for resection.

These criteria will ensure the probability of finding polyps during the explorations.

All the patients will give written informed consent.

Exclusion Criteria:

* Patients at a high risk of having major complications as perforation or hemorrhage, suspected or proven lower gastrointestinal bleeding, non-correctable coagulopathy or anticoagulant/clopidogrel therapy during procedure, inadequate bowel cleansing.
* ASA-IV patients.
* Urgent colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Number of polyps | During the procedure.
  With MiWEndo assisted colonoscopy, detect at least one polyp before colonoscopy in 10% of patients.
Number of adverse events. | During the procedure and up to 2 weeks after.
  Number of adverse events related with the use of the MiWEndo using the lexicon proposed by the American Society of Gastrointestinal Endoscopy (ASGE) (Cotton PB et al. GIE 2010;71:446-54).
Number of mural injuries. | During the procedure and up to 2 weeks after.
  Mural injuries related with the use of the MiWEndo.

SECONDARY OUTCOMES:
Number and size (adenomas and polyps). | During procedure.
  The number and size of all lesions (adenomas and all polyps) detected with MiWEndo-assisted colonoscopy.
True positives (TP), False positives (FP), False negatives (FN). | During procedure.
  The concordance with the lesions detected by the standard colonoscopy (TP, FP, FN).
Patients' comfort. | Immediately after the procedure and 2 weeks after.
  Patients' feedback related to colonoscopy using the Gloucester comfort score that ranges from 1 (no discomfort) to 5 (severe discomfort).
Perception of difficulty. | Immediately after the procedure.
  Perception of difficulty by the endoscopist based on a 5-points Likert scale (very easy to very difficult or very much to very little).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain